CLINICAL TRIAL: NCT03194568
Title: Safety and Feasibility of a Vertebral Body Tethering Technique for Pediatric Idiopathic Scoliosis
Brief Title: Vertebral Body Tethering Outcomes for Pediatric Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Cahill, MD (Other)
Responsible Party: Sponsor-Investigator, Patrick Cahill, MD, Attending Orthopaedic Surgeon, Children's Hospital of Philadelphia
Organization: Children's Hospital of Philadelphia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 17-013694
Record Dates: First submitted 2017-06-12; First posted 2017-06-21 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Idiopathic Scoliosis
Keywords: Scoliosis; Idiopathic Scoliosis; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Anterior Vertebral Tethering (Experimental): Subjects receiving Anterior Vertebral Tethering intervention.
  Interventions: Device: Anterior Vertebral Tether

INTERVENTIONS:
Device: Anterior Vertebral Tether — Vertebral body tethering through anterior thoracoscopic approach under general anesthesia and fluoroscopic guidance.

SUMMARY:
This study will assess whether Anterior Vertebral Tethering is a safe and feasible method of anterior approach surgery for spinal deformity in pediatric idiopathic scoliosis.

DETAILED DESCRIPTION:
Scoliosis is a condition in which the spine is deformed by a curvature in the coronal plane. It is generally associated with a twisting (axial plane) deformity as well. It can have a variety of underlying etiologies and the etiology is used to classify the types of scoliosis. Idiopathic scoliosis is sub-classified in two ways: by age of onset and by magnitude of deformity. Curves between 10 and 25 degrees are considered mild. Curves between 25 and 50 degrees are classified as moderate. Curves greater than 50 degrees are termed severe. The current standard of care for moderate scoliosis in patients with remaining growth is to utilize a thoracolumbosacral orthosis (TLSO brace) to prevent progression of deformity. The scientific evidence has supported the efficacy of this intervention in avoiding progression of the Cobb angle to 50 degrees or more.

If treated with a TLSO brace, many idiopathic scoliosis patients would conceivably be subjected to years of brace wear and the cost and psychological factors inherent therein. Additional downsides of brace treatment include the potentially negative psychosocial impact of wearing an external sign of deformity during adolescence, a key period of emotional development. Prior research has identified negative psychosocial effects related to wearing a brace in children.

Recent evidence has suggested that certain curve patterns will likely progress to 50 degrees or more, despite treatment with a TLSO brace. Sanders, et al. demonstrated a correlation of Cobb angle (greater than 35 degrees) and skeletal maturity (bone age 4 or less) to the risk of progression to 50 degrees or more, despite TLSO bracing. The evidence supports that the current practice of TLSO bracing is not an effective treatment to avoid progression to 50 degrees in these patients. It is on this population (thoracic Cobb angle greater than 35 degrees, bone age of 4 or less) that we intend to test the safety and feasibility of Anterior Vertebral Body Tethering to avoid curve progression to 50 degrees.

The study intervention is surgical orthopedic implantation of the Anterior Vertebral Tether Device, by way of thoracoscopic surgery under general anesthesia. The primary outcome measures include assessments of safety of the insertion procedure and of the device, as well as the secondary measure of feasibility by determining the ability to successfully implant the investigational device.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 8 to 16 years old at time of enrollment (inclusive)
2. Diagnosis of idiopathic scoliosis
3. Sanders bone age of less than or equal to 4
4. Thoracic curve of greater than or equal to 35 degrees and less than or equal to 60 degrees
5. Lumbar curve less than 35 degrees
6. Patient has already been identified for and recommended to have surgical intervention
7. Spina bifida occulta is permitted
8. Spondylolysis or Spondylolisthesis is permitted, as long as it is non-operative, the subject has not had any previous surgery for this, and no surgery is planned in the future

Exclusion Criteria:

1. Pregnancy (current)
2. Prior spinal or chest surgery
3. MRI abnormalities (including syrinx greater than 4mm, Chiari malformation, or tethered cord)
4. Neuromuscular, thoracogenic, cardiogenic scoliosis, or any other non-idiopathic scoliosis
5. Associated syndrome, including Marfan syndrome or neurofibromatosis
6. Sanders bone age greater than 4
7. Thoracic curve less than 35 degrees or greater than 60 degrees
8. Lumbar curve greater than or equal to 35 degrees
9. Unable or unwilling to firmly commit to returning for required follow-up visits
10. Investigator judgement that the subject/family may not be a candidate for the intervention

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Cahill, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Anterior Vertebral Tethering
Started | 20
Completed | 16
Not Completed | 4
Not completed — Withdrawn due to need for re-operation related to an anticipated device SAE | 4

BASELINE CHARACTERISTICS:
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 12 (1.94)
Age, Customized [Median (Standard Deviation); unit: years]
  Age at first diagnosis of Idiopathic Scoliosis | 9 (2.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20
Menarche status [Count of Participants; unit: Participants]
  Yes | 6
  No | 10
  N/A, Male | 4
Height (cm) [Median (Standard Deviation); unit: cm] | 159.4 (12.43)
Weight (kg) [Median (Standard Deviation); unit: kg] | 45.8 (13.82)
Degree of thoracic rib hump [Median (Standard Deviation); unit: Degrees] — Data collected using a scoliometer
  Degrees | 13 (4.64)
Thoracic Rib Hump Side [Count of Participants; unit: Participants]
  Right | 20
  Left | 0
Degree of lumbar rib hump [Median (Standard Deviation); unit: Degrees] — Data collected using a scoliometer
  Degrees | 6 (2.72)
Lumbar rib hump side [Count of Participants; unit: Participants]
  Left | 20
  Right | 0
Coronal Thoracic Cobb Angle [Median (Standard Deviation); unit: Degrees] | 51.5 (7.25)
Coronal Lumbar Cobb Angle [Median (Standard Deviation); unit: Degrees] | 29 (6.77)
Bending Thoracic Cobb Angle [Median (Standard Deviation); unit: Degrees] | 20.5 (10.56)
Bending Lumbar Cobb Angle [Median (Standard Deviation); unit: Degrees] — Population: Lumbar bending X-Ray not taken for 1 subject at baseline
  Degrees
    number analyzed (Participants) | 19
    (all) | 5 (9.83)
Sanders Bone Age [Count of Participants; unit: Participants] — Based on a scale of 0-8, the Sanders maturity scale considers level 0 to be slow growth in early adolescence whereas 8 is categorized as full skeletal maturity
  Participants
    0 | 0
    1 | 0
    2 | 2
    3 | 10
    4 | 8
    5 | 0
    6 | 0
    7 | 0
    8 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Intra-operative and post-intervention medical events or signs and symptoms of complications arising after the start of study intervention will be captured. The event description, date of onset, end date, severity, and outcome will be documented. The frequencies, type, body system, severity, and relationship to the study intervention will also be summarized. A distinction will be made between those events which are "device-related" and "non device-related".
Time Frame: up to 2 years
Population: Four of the subjects were withdrawn from the study prior to the 2 year completion date due to need for re-operation related to an anticipated device SAE. All data reported for these subjects were obtained prior to withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 20
Participants
  Subjects that experienced a device-related AE | 11
  Subjects that experienced a device-related SAE | 7
  Subjects that experienced a non-device related AE | 20
  Subjects that experienced a non-device related SAE | 0

2. Secondary Outcome: Comparison of Pre-Operative and Post-Operative Cobb Angle
Description: The exploratory therapeutic endpoint used for feasibility will be change in post-operative Cobb angle compared to pre-operative Cobb angle, measured on coronal radiograph of the spine.
Time Frame: up to 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 20
Participants
  Thoracic curve <50° without a secondary spinal fusion or other revision surgery | 14
  Thoracic curve >50°, or requiring a secondary spinal fusion or other revision surgery | 6

3. Secondary Outcome: Comparison of Pre-Operative and Post-Operative SRS 30 Scores
Description: The Scoliosis Research Society 30 (SRS-30) questionnaire will be administered at pre-operative and post-operative time points. This questionnaire measures health-related quality of life outcomes. It consists of 30 questions divided into five domains: Function/Activity (5 questions), Pain (5 questions), Self-image/Appearance (5 questions), Mental Health (5 questions), and Satisfaction with management (2 questions). The remaining 8 questions are a combination of different domains. Each question is scored on a 5-point scale (1 = worst, 5 = best). To score each domain, sum the scores of the questions within that domain and then divide by the number of questions in that domain to get an average score. To calculate the total overall score, sum all the individual question scores and then divide by the total number of questions (30). Higher scores indicate better health-related quality of life.
Time Frame: up to 2 years
Population: Four of the 20 initial subjects were withdrawn from the study prior to final follow-up administration of SRS questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Anterior Vertebral Tethering
Number analyzed (Participants) | 20
score on a scale
  Pre-operative Function/Activity | 4.4 (0.4)
  Pre-operative Pain | 4.3 (0.7)
  Pre-operative Self-image/Appearance | 3.6 (0.8)
  Pre-operative Mental Health | 4.2 (0.6)
  Pre-operative Satisfaction with management | 3.5 (0.9)
  Pre-operative total score | 4.1 (0.5)
  Post-operative Function/Activity: number analyzed (Participants) | 15
  Post-operative Function/Activity | 4.5 (0.4)
  Post-operative Pain: number analyzed (Participants) | 15
  Post-operative Pain | 4.6 (0.5)
  Post-operative Self-image/Appearance: number analyzed (Participants) | 15
  Post-operative Self-image/Appearance | 4.2 (0.7)
  Post-operative Mental Health: number analyzed (Participants) | 15
  Post-operative Mental Health | 4.1 (0.7)
  Post-operative Satisfaction with management: number analyzed (Participants) | 15
  Post-operative Satisfaction with management | 4.2 (1.0)
  Post-operative total score: number analyzed (Participants) | 15
  Post-operative total score | 4.3 (0.5)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected up to 2 years after the date of surgical implant for each subject. Additionally, the majority of the subjects enrolled in this study have also enrolled in an observational long-term follow up study.
Description: Surgery and Post-operative Phase (Day 0 - POD 90): All AEs & SAEs will be noted.
  Extended Follow-up (POD 91-POD 730): All SAEs recorded. Only AEs which are deemed "device related" recorded.
  Long-term Follow-Up (POD 730 through two years after skeletal maturity): All SAEs identified from the medical records that are considered device related, up to two years after skeletal maturity, will be reported in accordance with FDA requirements. This will be performed under a separate research protocol.
Arm/Group | Anterior Vertebral Tethering
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anterior Vertebral Tethering (N=20)
Grade IIIB (Injury, poisoning and procedural complications) | 6 — Requiring surgical, endoscopic or radiological intervention under general anesthesia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Vertebral Tethering (N=20)
Grade I (Respiratory, thoracic and mediastinal disorders) | 20 (56) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade II (Injury, poisoning and procedural complications) | 1 (1) — Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions and total parenteral nutrition are also included.
Grade I (Gastrointestinal disorders) | 12 (16) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade I (Skin and subcutaneous tissue disorders) | 6 (7) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade I (Musculoskeletal and connective tissue disorders) | 16 (52) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade I (General disorders) | 3 (4) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade I (Cardiac disorders) | 1 (1) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade I (Psychiatric disorders) | 1 (1) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.
Grade I (Product Issues) | 3 (3) — Deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions. Also includes wound infections opened at the bedside.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03194568/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT03194568/ICF_001.pdf